CLINICAL TRIAL: NCT04010721
Title: Effects of Parameters of the Electrical Stimulation on Loudness in Oticon Medical Cochlear Implant Patients. Investigational Study for Cochlear Implant Fitting Facilitation
Brief Title: Effects of Pulses on Loudness
Acronym: EfPuL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PIC-19
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss, Cochlear
Keywords: Cochlear implant
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental : experiment 1,2 and 3 (Other): One user included participates all experiments:
  * Visit 1 : experiment 1
  * Visit 2 : experiment 2
  * Visit 3 : experiment 3
  Interventions: Device: Experiment 1; Device: Experiment 2:; Device: Experiment 3

INTERVENTIONS:
Device: Experiment 1 — Stimulation of one electrode at a time
Device: Experiment 2: — Stimulation in groups of 4, 8 and 12 electrodes
Device: Experiment 3 — Stimulation total duration from 10 to 600 ms

SUMMARY:
The aim of this study is to investigate the effect of varying additional factors on loudness summation in Neuro Zti Cochlear Implant users.

DETAILED DESCRIPTION:
Primary objective:

- To assess the effect of the number and spatial distribution of active electrodes on the stimulation charge required to achieve the loudness associated with C and T levels (Experiment 2).

Secondary objectives:

* To assess how loudness is affected by changes in electrical charge of individual pulses made by adjusting the pulse amplitude versus adjusting pulse duration (Experiment 1).
* To assess how loudness elicited by a train of pulses is affected by the duration of that pulse train (Experiment 3).

Experiment 1:

The test will investigate the effect of loudness on changes in electrical charge of individual pulses, made by separately adjusting pulse amplitude or pulse width. The electrical charge required to elicit different loudness ("just-audible", "soft", "medium", "comfortable", "loud but comfortable") either when increasing the amplitude or the duration of the pulses.

Experiment 2:

The test will investigate the effect of the number of stimulating electrodes and their distribution within the cochlea on the stimulation levels required to achieve T-levels and C-levels and to elicit different loudness ("just-audible", "soft", "medium", "comfortable", "loud but comfortable").

Experiment 3:

The test will investigate the effect on loudness of trains of pulses elicited by modifications to the duration of those trains, when operating around T and C levels. Stimulation durations ranging from 10 to 600 ms will be tested. Pulse trains will be presented to either one or several electrodes to elicit different loudness ("just-audible", "soft", "medium", "comfortable", "loud but comfortable").

ELIGIBILITY:
Inclusion Criteria:

* Neuro One or Neuro 2 user
* Unilateral or bilateral recipient
* 12 months CI experience to allow for acclimatization to the CI sound processing and pathological changes that could alter the electrode - tissue interface and therefore T- & C-levels.
* Having at least 7 step sizes on three electrodes in their current clinical map (for experimentation 1).
* Able and willing to provide reliable threshold and comfort level judgements

Exclusion Criteria:

* Medical conditions that contraindicate the study tests (e.g. tinnitus, dizziness)
* Unrealistic expectations from the candidate regarding the possible benefits, risks, and limitations that are inherent to the device
* Unwillingness or inability of the candidate to comply with all investigational requirements
* Vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Experiment 2: the effect of number of electrodes on loudness | 2 hours
  Changes in electrical charge (nC) needed to achieve C-level and T-level. The charge is the results of Intensity*Duration of a pulse, in µA and µs respectivelly. If either the amplitude or the duration of the pulse is modified, the charge will be modified as well.

SECONDARY OUTCOMES:
Experiment 1 : the effect of pulse amplitude and pulse duration on loudness | 2 hours
  Change of the charge (nC) required to elicit different loudness. The charge is the results of Intensity*Duration of a pulse, in µA and µs respectivelly. If either the amplitude or the duration of the pulse is modified, the charge will be modified as well.
Experiment 3 : the effect of stimulation duration on loudness | 2 hours
  Change of the charge (nC) to elicit th most comfortable loudness (C-level). The charge is the results of Intensity*Duration of a pulse, in µA and µs respectivelly. If either the amplitude or the duration of the pulse is modified, the charge will be modified as well.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe VINCENT, Principal Investigator — CHRU LILLE
Locations (1):
- CHU Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No